CLINICAL TRIAL: NCT04347941
Title: Awake Prone Positioning to Reduce Invasive VEntilation in COVID-19 Induced Acute Respiratory failurE
Acronym: APPROVE-CARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment for trial was terminated on January 26, 2021 after a third interim analysis demonstrated that a pre-defined statistical criteria for efficacy were met as part of meta-trial study of awake prone positioning.
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor, Anaesthesia and Intensive Care Medicine, School of Medicine, NUI Galway, University College Hospital Galway
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPROVE-CARE-2020
Record Dates: First submitted 2020-04-08; First posted 2020-04-15 (Actual); Results first posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: ARDS, Human; Mechanical Ventilation Complication; COVID19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — Prone Position; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone Positioning (Experimental): Intervention patients will remain up to 16 hours per day in Prone Positioning with 45 minutes breaks for meals
  Interventions: Procedure: Prone Positioning
- Standard Care (Active Comparator): Control patients will receive full standard care. Prone Positioning as a rescue intervention is permitted and is recorded.
  Interventions: Procedure: Standard of care.

INTERVENTIONS:
Procedure: Prone Positioning — Patient will be asked to remain for at least one hour and to a maximum total of 16 hours in prone position with 45 minutes breaks for meals. Immediately prior to proning, if spO2 <94% on FiO2 0.4, start on 100% O2 to ensure stability during proning. A nurse or assistant will assist patient to turn on side and then face down with the support of pillows as required for comfort, ensure that they are predominantly on their chest rather than on their side. Arms can be at side, in swimmer position and can be moved to patients' comfort, pillows under knees and chest for comfort and call bell to be at patient's arm's length. Vitals and work of breathing score will be measured before and at 1 hour into each proning session and at the end of each session. Total length of time in prone position will be recorded. Intervention to continue daily until oxygen requirement to maintain spO2 >94% is below FiO2 0.4 via venturi facemask or high flow nasal cannula
  Arms: Prone Positioning
Procedure: Standard of care. — Standard of care. Prone positioning may be administered as a rescue therapy
  Arms: Standard Care

SUMMARY:
Prone positioning (PP) is an effective first-line intervention to treat moderate-severe acute respiratory distress syndrome (ARDS) patients receiving invasive mechanical ventilation, as it improves gas exchanges and lowers mortality.The use of PP in awake self-ventilating patients with (e.g. COVID-19 induced) ARDS could improve gas exchange and reduce the need for invasive mechanical ventilation, but has not been studied outside of case series.The investigators will conduct a randomized controlled study of patients with COVID-19 induced respiratory failure to determine if prone positioning reduces the need for mechanical ventilation compared to standard management.

DETAILED DESCRIPTION:
Prone positioning (PP) is an adjunctive therapy used that has been proven to save lives in sedated patients with confirmed moderate-severe acute respiratory distress syndrome (ARDS) receiving invasive mechanical ventilation (MV). PP involves placing patients in the prone, i.e. face down position for time periods of up to 16 hours per day. PP promotes lung homogeneity, improves gas exchange and respiratory mechanics permitting reduction of ventilation intensity, and reducing ventilator-induced lung injury (VILI).

Maintaining self-ventilation is associated with increased aeration of dependent lung regions, less need for sedation, improved cardiac filling and removes the risk of VILI, and so is an important therapeutic goal in hypoxic patients. The use of PP in awake self-ventilating patients with COVID-19 induced acute hypoxic respiratory failure (AHRF) and/or ARDS could improve gas exchange and reduce the need for invasive MV, but has not been studied outside of case series.

However, an increase in oxygenation does not necessarily reduce the risk of invasive MV. PP has significant attached risks such as causing pressure sores in patients, PP is uncomfortable for some patients, it increases nursing workload, and if ineffective could hinder the delivery of other (effective) medical care. Hence there is a need to determine if PP of awake patients is effective in reducing the need for invasive MV. This multi-centre, open label, randomized controlled study of COVID-19 induced AHRF/ARDS will determine if PP reduces the need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed COVID19 infection
* Bilateral Infiltrates on CXR
* SpO2 <94% on FiO2 40% by either venturi facemask or high flow nasal cannula
* RR <40
* Written informed consent

Exclusion Criteria:

* Age <18
* Uncooperative or likely to be unable to lie on abdomen for 16 hours
* Receiving comfort care only
* Multi-organ failure
* RR>40
* Contraindication to PP (e.g. vomiting, abdominal wound, unstable pelvic/spinal lesions, pregnancy >20/40 gestation, severe brain injury).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Galway University Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Electronic Case report form following informed consent, all patient identification removed, and individual patient response to intervention will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: up to 15 years post study

REFERENCES:
- [Background] Ehrmann S, Li J, Ibarra-Estrada M, Perez Y, Pavlov I, McNicholas B, Roca O, Mirza S, Vines D, Garcia-Salcido R, Aguirre-Avalos G, Trump MW, Nay MA, Dellamonica J, Nseir S, Mogri I, Cosgrave D, Jayaraman D, Masclans JR, Laffey JG, Tavernier E; Awake Prone Positioning Meta-Trial Group. Awake prone positioning for COVID-19 acute hypoxaemic respiratory failure: a randomised, controlled, multinational, open-label meta-trial. Lancet Respir Med. 2021 Dec;9(12):1387-1395. doi: 10.1016/S2213-2600(21)00356-8. Epub 2021 Aug 20. PMID 34425070
- [Result] Tavernier E, McNicholas B, Pavlov I, Roca O, Perez Y, Laffey J, Mirza S, Cosgrave D, Vines D, Frat JP, Ehrmann S, Li J. Awake prone positioning of hypoxaemic patients with COVID-19: protocol for a randomised controlled open-label superiority meta-trial. BMJ Open. 2020 Nov 11;10(11):e041520. doi: 10.1136/bmjopen-2020-041520. PMID 33177145
- See also: Result of Meta-trial in which RCT was incorporated — https://doi.org/10.1016/S2213-2600(21)00356-8

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prone Positioning | Standard Care
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with suspected or confirmed COVID-19 pneumonia requiring high flow nasal cannula oxygen were randomized to either awake prone positioning or standard of care. The primary outcome was the requirement for invasive mechanical or death post 28 days randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prone Positioning | Standard Care | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Ireland | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Prone Positioning on Requirement for Invasive Mechanical Ventilation or Death in Patients With COVID 19 Induced Respiratory Failure.
Description: A measure of effect of awake prone positioning in patients with confirmed or suspected COVID-19 acute hypoxemic respiratory failure undergoing supplemental oxygen via high flow nasal cannular oxygen on reducing requirement for invasive mechanical ventilation or death. Outcome measure is calculated as a count of the number of patients who went onto require invasive mechanical ventilation or died up to 28 days post randomization.
Time Frame: Up to 28 days post randomisation
Population: Number of patients who required invasive mechanical ventilation or who died in each group up to 28 days post randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Prone Positioning | Standard Care
Number analyzed (Participants) | 12 | 12
Participants | 0 | 2

2. Secondary Outcome: Length of Time Tolerating Prone Positioning
Description: description of duration of prone positioning in hours per day from day 0 to day 14 in trial
Time Frame: Daily during intervention up to 14 days post randomisation
Population: description of duration of prone positioning in hours per day from day 0 to day 14 in trial
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prone Positioning | Standard Care
Number analyzed (Participants) | 12 | 12
hours | 3.3 (2.7) | 1.0 (2.5)

3. Secondary Outcome: PaO2/FiO2 Ratio Measured Before Prone Positioning
Description: Measure of change in oxygenation before intervention in the patients assigned to awake prone positioning
Time Frame: Immediately before intervention
Population: paO2 to fiO2 ratio before prone positioning in the group assigned to undergo awake prone positioning
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Standard of Care: Patients with suspected or confirmed COVID-19 pneumonia who are randomized to not undergo awake prone positioning but receive otherwise identical care as the awake prone positioning group.
Arm/Group | Prone Positioning | Standard of Care
Number analyzed (Participants) | 12 | 12
ratio | 144 (52) | 114 (40)

4. Secondary Outcome: PaO2/FiO2 Ratio After 1 Hours of Prone Positioning
Description: Measure of change in oxygenation following patients being placed in the prone position for 1 hour
Time Frame: During intervention
Population: change in paO2 one hour after proning in the individuals who were in the intervention group and underwent awake prone positioning
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Prone Positioning
Number analyzed (Participants) | 12
ratio | 33 (32)

5. Secondary Outcome: SpO2/FiO2 Ratio Measured Before Prone Positioning
Description: Measure of oxygenation using pulse oximetry before intervention where ABG not available
Time Frame: Immediately before intervention
Population: spO2 to fiO2 ratio at baseline prior to awake prone position in those undergoing awake prone position, and on the morning post enrolment for patients undergoing standard of care treatment
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Standard of Care: Patients with suspected or confirmed COVID-19 pneumonia requiring high flow nasal cannula oxygen who were randomized to not undergo awake prone positioning as part of their management and received otherwise identical treatment as the awake prone positioning arm.
Arm/Group | Prone Positioning | Standard of Care
Number analyzed (Participants) | 12 | 12
ratio | 193 (45) | 178 (52)

6. Secondary Outcome: SpO2/FiO2 Ratio After 1 Hour in Prone Positioning
Description: Measure of oxygenation 1 hour after intervention where ABG not available
Time Frame: During Intervention
Population: spO2 to fiO2 ratio following 1 hour in prone position
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Prone Positioning
Number analyzed (Participants) | 12
ratio | 247 (53)

7. Secondary Outcome: Number Requiring Increase in Ventilatory Assistance
Description: Number of patients in each group requiring an increase in the respiratory support from baseline high flow nasal cannula oxygen post randomization up to 28 days later, defined as need for continuous positive airway pressure (CPAP), bilevel positive airway pressure (biPAP)
Time Frame: Up to 28 days post randomisation
Population: Number of patients in each group requiring an increase in the respiratory support from baseline high flow nasal cannula oxygen post randomization up to 28 days later, defined as need for continuous positive airway pressure (CPAP), bilevel positive airway pressure (biPAP)
Measure: Count of Participants; unit: Participants
Arm/Group | Prone Positioning | Standard Care
Number analyzed (Participants) | 12 | 12
Participants | 4 | 4

8. Secondary Outcome: Work of Breathing Assessment (Respiratory Distress Scale)
Description: Measure of work of breathing in COVID-19 based on Oxygen Delivery Device, Oxygen Saturation and respiratory rate and accessory muscle use with 0-3 Mild, 4-6 Moderate and 7-10 Severe
Time Frame: Immediately before and during intervention
Population: We did not carry out this aspect of the study due to constraints related to the Pandemic
Arm/Group | Prone Positioning | Standard Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Changes in Bioimpedance Measures of Lung Edema in Patients in PP
Description: Substudy examining use of bioimpedance as a surrogate measure of lung edema following prone positioning
Time Frame: During intervention
Population: Due to constraints related to the pandemic, this aspect of the study was not carried out.
Arm/Group | Prone Positioning | Standard Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Use of Awake Prone Positioning as a Rescue Intervention in Control Patients
Description: Number of patients who underwent rescue awake prone positioning in control patients by physicians in response to hypoxia
Time Frame: Up to 28 days post randomisation
Population: Number of patients who underwent awake prone positioning in the control arm of the study as a rescue manoeuvre in response to hypoxia.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: hospital discharge or 28 days
Arm/Group | Prone Positioning | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Study was terminated after an interim analysis of a prospective meta-trial in which the patients reached statistical criteria for efficiency

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT04347941/Prot_SAP_000.pdf